CLINICAL TRIAL: NCT01817413
Title: Revascularisation Versus Mineral Trioxide Aggregate in the Management of Non-Vital Immature Permanent Incisors in a Young Population: A Randomised Controlled Trial (Pilot Study)
Brief Title: Comparison of Two Dental Techniques Used to Treat Teeth Which Have Become Infected or Painful Following Trauma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Laura Gartshore, Clinical Lecturer & Postgraduate Research Student, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD&I 3968, UoL000590; Controlled Trials (Registry Identifier: ISRCTN34934882)
Record Dates: First submitted 2013-03-18; First posted 2013-03-25 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Apexification; Apexogenesis; Pulp Necrosis; MTA; Pulp Revascularisation; Periapical Periodontitis; Non-vital Immature Tooth
Keywords: Calcium hydroxide; Pulp regeneration; Regenerative endodontics; Pulp revitalisation; Triple antibiotic paste; Root canal therapy; Root end closure; Tooth root; Tooth apex; Dental trauma; Non-vital; Immature; Incisor; Periapical periodontitis; Dental pulp
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis | interventions — mineral trioxide aggregate; Pemetrexed; Apexification; Regenerative Endodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apexification with MTA (Active Comparator): The control group will receive:
  Visit 1: root canal dressing with calcium hydroxide Visit 2: apexification with mineral trioxide aggregate (MTA), followed by obturation of the root canal with gutta percha.
  Treatment will be carried out over two visits, two weeks apart.
  Interventions: Procedure: Mineral trioxide aggregate
- Pulp revascularisation (Experimental): The experimental group will receive:
  Visit 1: root canal dressing with triple antibiotic paste Visit 2: pulp revascularisation procedure Treatment will be carried out over two visits, two weeks apart.
  Interventions: Procedure: Revascularisation

INTERVENTIONS:
Procedure: Mineral trioxide aggregate — An apical barrier of mineral trioxide aggregate (MTA cement) will be placed in the tooth root at the open apex in order to achieve root end closure via an apexification technique
  Other Names: MTA; MTA cement; Apexification
  Arms: Apexification with MTA
Procedure: Revascularisation — Pulp revascularisation will be induced by instrumentation through the open apex so that a blood clot forms within the root canal in order to achieve root end closure via apexogenesis
  Other Names: Regenerative endodontics; Pulp revitalisation; Apexogenesis
  Arms: Pulp revascularisation

SUMMARY:
Children often damage their front teeth. In approximately 6% of cases, the nerve inside the affected tooth dies (becomes 'non-vital') and natural root development stops. In these cases, the tooth requires a root canal treatment in order to prevent problems such as pain and dental abscesses from arising. However, because the roots of these young teeth are not fully formed, they are weaker and prone to fracture. In addition, root canal treatment is difficult because a root canal filling cannot be placed in a tooth which is not yet fully formed, due to the fact that the root has an 'open' end.

To enable root canal treatment to be carried out, a 'barrier' must be placed at the end of the 'open' root. This can be done using materials called Calcium Hydroxide or Mineral Trioxide Aggregate (MTA). These materials are placed inside the root and sealed into the tooth. However, although they help to provide a barrier, they do not help to strengthen the walls of the root. Treatment with these materials requires multiple visits to the dentist, over a period of up to 18 months.

There is evidence to suggest that an alternative treatment involving 'revascularisation' (recovery of the blood supply to the tooth) and the use of a triple antibiotic paste allows 'natural' root growth to restart, and also strengthens the walls of the root. Treatment can often be carried out in just two visits.

The aim of this study is to discover whether there is a difference between one of two methods of treating non-vital teeth with open ends. It is thought that there will be no significant differences seen between the results of the two techniques.

Children with teeth that fall into this category and require root canal treatment will be given one of two treatments, both of which aim to treat infection, close the root end and to allow healing to take place.

Teeth will receive one of the following methods of root treatment:

1. Revascularisation (recovery of the natural blood supply to the tooth) following placement of an antibiotic paste into the tooth root. The aim of this treatment is to allow 'natural' root growth to restart. Root growth will allow the tooth to form at barrier at the end of the root. No root canal filling will then be necessary.
2. Closure of the open root end by placement of an artificial barrier at the end of the root so that a root canal filling can then be placed. This will be done with a dental material called Mineral Trioxide Aggregate (MTA). Non-vital teeth with an open end are routinely treated in this way at Liverpool Dental Hospital.

DETAILED DESCRIPTION:
Participants will be randomly allocated in to one of the above treatment groups. This means that neither the participants, nor the researchers, will be able to choose which group a participant will be allocated to.

In both techniques, in order to learn about the bacteria involved in non-vital teeth, the investigators will take samples of the bacteria within the root canal.

The outcomes of the study will provide us with further information about root growth, the bacteria involved in infection of non-vital teeth and the success of the different treatment methods that are available. This information will enable us to increase our understanding of the treatment of non-vital teeth with an open end and help us to explain our treatments to future patients.

All children presenting to Liverpool University Dental Hospital aged between 7 and 25 years of age and who are medically well and cooperative to receive prolonged treatment in the dental chair are eligible to take part in the study if they have a damaged upper front adult tooth in which the nerve has died and the root is open ended. Unfortunately, if there is dental decay in the tooth or a fracture of the root then these teeth are not suitable for this study. In some cases following damage to a tooth, the root of the tooth starts to dissolve and unfortunately these teeth are also not suitable for this study.

Suitable patients attend with their parent or carer for a consultation to the Paediatric Dentistry Clinic at Liverpool University Dental Hospital. Following this visit, if a suitable patient wishes to join our study the investigators will arrange two further visits during which the dental treatment will take place. Following completion of treatment, patients will be asked to return for four check ups over the next year so that the investigators can check that they are happy and that treatment has been successful.

There are no risks or disadvantages to taking part in this study. However, if the tooth does not respond to treatment, or if symptoms of infection arise, then alternative treatment methods may be initiated as necessary.

The study is being funded by the Royal Liverpool and Broadgreen University Hospitals NHS Trust and by the University of Liverpool.

ELIGIBILITY:
Inclusion Criteria for participants:

* Between 7 and 25 years of age
* Have no significant medical history
* Cooperative in the dental chair
* Able to commit to the recall schedules prescribed by the study
* Have one or more traumatised non-vital permanent maxillary central incisors with incomplete root development

Exclusion Criteria for participants:

* Have a medical history that may complicate treatment
* Have a medical history for which the study procedures may place the patient at increased risk
* Have a diagnosis of avulsion or severe intrusion following dental trauma

Exclusion Criteria for Permanent maxillary central incisors:

* Less than half formed
* Have anatomical complexity (such as dens invaginatus)
* Have horizontal or vertical root fractures present
* Have evidence of root resorption

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evidence of periapical healing | 12 months
  Teeth will be reviewed clinically and radiographically at 3, 6, 9 and 12 months in order to monitor healing progress.
  Final outcome measures will be recorded at 12 months.
Presence of a satisfactory apical barrier | 12 months
  Teeth will be reviewed clinically and radiographically at 3, 6, 9 and 12 months in order to monitor healing progress.
  Final outcome measures will be recorded at 12 months.

SECONDARY OUTCOMES:
Patient satisfaction | 12 months
  Teeth will be reviewed clinically and radiographically at 3, 6, 9 and 12 months in order to monitor healing progress.
  Final outcome measures will be recorded at 12 months.
Evidence of root development | 12 months
  Teeth will be reviewed clinically and radiographically at 3, 6, 9 and 12 months in order to monitor healing progress.
  Final outcome measures will be recorded at 12 months.
A satisfactorily restored tooth | 12 months
  Teeth will be reviewed clinically and radiographically at 3, 6, 9 and 12 months in order to monitor healing progress.
  Final outcome measures will be recorded at 12 months.
Absence of signs and symptoms of failure of treatment (pain, mobility, tenderness to percussion, pathology e.g.sinus or swelling) | 12 months
  Teeth will be reviewed clinically and radiographically at 3, 6, 9 and 12 months in order to monitor healing progress.
  Final outcome measures will be recorded at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: C C Youngson, Study Chair — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

REFERENCES:
- See also: Current Controlled Trials Registration — http://www.controlled-trials.com/ISRCTN34934882